CLINICAL TRIAL: NCT01070485
Title: An Open-label Phase IIa, Non-randomized Study of Alpharadin® in Breast Cancer Patients With Bone Dominant Disease no Longer Considered Suitable for Endocrine Therapy
Brief Title: BAY88-8223, Alpharadin, Breast Cancer Patients With Bone Dominant Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15468; 2009-012189-30 (EudraCT Number); BC1-09 (Other: Algeta ASA)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer; Bone Metastases
MeSH Terms: conditions — Breast Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium-223 dichloride (Xofigo, BAY 88-8223) (Experimental): Patients were to receive 4 intravenous administrations of Radium-223 at a dose of 50 kBq/kg body weight (b.w) at intervals of 4 weeks. Radium-223 was given as add-on therapy to existing bisphosphonate therapy.
  Interventions: Drug: Radium-223 chloride (BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 chloride (BAY88-8223) — The required volume of study drug to be administered to a patient was calculated using the patient's body weight (50 kBq/kg b.w.).

SUMMARY:
The purpose of the study is to investigate if multiple (up to four) intravenous injections of Xofigo (Alpharadin) have any clinically relevant effect on bone markers in breast cancer patients with bone dominant disease who have progressed on endocrine therapy and are no longer considered suitable for endocrine therapy. In addition the safety of Xofigo (Alpharadin) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is female, and either post-menopausal (cessation of menses for more than 1 year) or surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy) or in therapy-induced premature menopause with LHRH agonists. If of childbearing potential the result of a urine human chorionic gonadotropin pregnancy test, performed on the same day as and with the result known before study drug administration, must be negative.
* Histological or cytological evidence of primary breast cancer.
* Bone dominant disease (with or without metastases in soft tissue, lymph nodes and/or skin) with at least one non-irradiated bone metastasis on planar bone scintigraphy/SPECT ± CT within previous the 12 weeks.
* Patient has unequivocally progressed on endocrine therapy and further benefit from endocrine therapy is considered unlikely (progression must be documented based on imaging and/or other clinically relevant information).
* Patient has been on bisphosphonate therapy for at least 3 months prior to treatment start and no change to bisphosphonate therapy is expected during the treatment phase of the study, or patient is not being treated with bisphosphonates, and such treatment is not planned to start during the treatment period.
* Latest endocrine therapy stopped at least 2 weeks prior to treatment start.
* ECOG PS 0 - 2.
* Life expectancy ≥6 months.
* Patient fulfils the following certain laboratory requirements.

Exclusion Criteria:

* Received an investigational drug within 4 weeks prior to the administration of Alpharadin, or is scheduled to receive one during the treatment period.
* Received chemotherapy, immunotherapy, or external beam radiation therapy within the last 4 weeks prior to administration of study drug, or has not recovered from acute ARs as a result of such therapy.
* Is likely to require chemotherapy or immunotherapy within the 16 weeks treatment period.
* Presence of imminent or established spinal cord compression based on clinical findings and/or MRI.
* Presence of other currently active (relapse within the last 3 years) malignancy (except non-melanoma skin cancer) that are not breast cancer metastases.
* Presence of unequivocal visceral metastases requiring chemotherapy treatment in the next 6 months, based on Investigator's judgement. Brain metastases are allowed only if well controlled and if not associated with symptoms. Treatment for brain metastasis should have been completed at least 8 weeks prior to treatment start.
* Patients with any other serious illness or medical condition, such as:

  * any uncontrolled infection
  * clinical heart failure severe enough to cause marked limitation of activity, and who is only comfortable at rest; or heart failure more severe than this (NYHA Heart Failure Class III or IV)
  * Crohn's disease or ulcerative colitis
  * Bone marrow myelodysplasia
  * Unmanageable faecal incontinence

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in bone markers (urine levels of NTX (uNTX) and bone-alkaline phosphatase (ALP) | 16 weeks

SECONDARY OUTCOMES:
All safety data, including adverse events, changes in laboratory variables, vitals signs, physical examination, late toxicity | 1 year
Biochemical markers (additional bone markers and CA15.3) | 16 weeks
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | 1 year
Pain | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Belgium (2):
  - Brussels
  - Liège
- Oslo, Norway
- Sheffield, United Kingdom